CLINICAL TRIAL: NCT06098807
Title: Family Centered Treatment for Problematic Gaming and Excessive Screen Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Emma Claesdotter-Knutsson, Associate Professor, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-05533-01
Record Dates: First submitted 2023-10-08; First posted 2023-10-25 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Internet Gaming Disorder; Internet Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Familiy Based Treatment (Experimental): ;one session per week during a period of four weeks with high quality content. The sessions will be performed at CAP location in Lund. The treatment will be performed by a clinician at CAP who could be a doctor, psychologist or health counselor - all with cognitive behavioral therapy competence. The sessions will be in group settings, separately for children and parents. In that sense, children will be included in a group with other children and parents will be included in a group with other parents. Each group will have 1-2 therapists leading the program. The theme of the week will be the same for both parent and child group, although the delivery will potentially differ. We expect that a session will last approximately 90 min with a 15-minute coffee break included.
  Interventions: Behavioral: Family Centered Treatment for Problematic Gaming and Excessive Screen Use

INTERVENTIONS:
Behavioral: Family Centered Treatment for Problematic Gaming and Excessive Screen Use — Based on earlier implementation research with parents and children the treatment is likely to consist of a low number of sessions ;one session per week during a period of four weeks with high quality content. The sessions will be performed at CAP location in Lund. The treatment will be performed by a clinician at CAP who could be a doctor, psychologist or health counselor - all with cognitive behavioral therapy competence. The sessions will be in group settings, separately for children and parents. In that sense, children will be included in a group with other children and parents will be included in a group with other parents. Each group will have 1-2 therapists leading the program. The theme of the week will be the same for both parent and child group, although the delivery will potentially differ. We expect that a session will last approximately 90 min with a 15-minute coffee break included.

SUMMARY:
The general increase in screen time as a time-consuming leisure activity among children and youth has been a puzzle to the adult world. Specifically, parents and professionals who work with children and youth express concern for the effect excessive screen time including gaming may have for child and youth development. The clinical picture of problematic gaming and excessive screen time describes compulsion, psychiatric and physical symptoms, impaired cognitive development, and school performance. The aim of this project is to set up and evaluate an easily accessible family centered treatment intervention for a child and adolescent psychiatry population. This study can lead to reduced suffering by optimization the care interventions for patients with problematic gaming and gambling.

DETAILED DESCRIPTION:
During the past 10 years, use of screen as in social media and video games has become one of the most common leisure activities for children and adolescents. According to the Swedish Internet Foundation, 94% of children in Sweden between ages 8 and 12 play internet games every day. Male and female screen behaviours and habits differ. Boys tend to play video games while girls are more active on social media. The general increase in screen time among children and youth, as a time-consuming leisure activity has been a puzzle to the adult world. Specifically, parents and professionals who work with children and youth express concern for the effect that screen time may have for child and youth development. Some research suggest that screen time in general and gaming in particular is an educational and skills training activity. Other research has concerns that video games can become a potentially pathological activity that interferes with everyday life with risks of developing psychiatric disorders such as internet gaming disorder (IGD). IGD is included in the Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5), as a condition necessitating further clinical experience and research before inclusion as a formal disorder. The WHO, on the other hand, has included Gaming Disorder in the International Classification of Diseases, eleventh revision (ICD-11), as a formal diagnosis. Experiencing addictive problems as a child may pose threat for future psychosocial development, including mental health and socioemotional development. In that sense, child and youth mental health services need to put more efforts into developing interventions that target children at risk to prevent the development of mental health problems among children and youth. To date, there are no evaluated preventive programs for child and youth with excessive screen time or problematic gaming in Sweden. Our research group from Lund University and Region Skåne, with Emma Claesdotter-Knutsson (E C-K) as a PI, has evaluated Relapse prevention (RP) as an individual treatment for problematic gaming in a Random Controlled trial (RCT) among children 12-18 years old in a Child and Adolescent Psychiatry (CAP) setting. This was one of the first treatment studies for children with problematic gaming in Europe. Although we discovered that the individual treatment of children and youth has promising effect on their gaming, we also found that that there were important pieces lacking when providing treatment for children with problematic gaming. The most prominent one was the lack of family, including parents, involvement in the treatment. Children and their development need to be seen from a system perspective - children develop in interaction with their environment/family. For children, parents are the closest socializing agents in their environment who with their parenting behaviours and practices pave the way for child developmental transitions. In that sense, the development of certain behaviours, such as gaming and excessive screen use may, at least to some extent, be related to family factors. It is then possible that child problematic screen time/gaming is not only attributed to the child itself, but to the family as a system. Therefore, we believe that parents need to be included in the preventive interventions targeting children and their families. Instead of only focusing on the child, changing the family environment, including parent-child interactions at home, may pose significant changes in the child's screen behaviour. This is a recognized logic from other family interventions such as Strengthening families program targeting families with children with behavioural problems and Cool Kids program targeting families with children with anxiety. In fact, parents whose children have undergone the RP-treatment in our project state that they need to and want to be involved in the child's treatment.

With this as a background, the overarching goal with this project is to develop and evaluate an easily accessible family program targeting children and adolescents with problematic gaming and excessive screen use.

ELIGIBILITY:
Inclusion criteria:

1. Age 12 to <18 years
2. Self-perceived problems in the family regarding computer gaming or screen use
3. Children/youth and guardians can read, write and communicate in Swedish
4. An available guardian who can participate in the treatment
5. Access to the internet
6. Possibility to participate in treatment sessions on site at the reception

Exclusion criteria:

1. Observed or suspected intellectual disability

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
SCREENS-Q | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  Screening form, for valuing children and adolescent´s screen time
GASA | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  Screening form, for diagnosis of computer game addiction
PARCA | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  (adapted) Screening form for assessing aspects of parent-child relationship and parenting practices
FCU | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  Five items measure parent-child warmth, and three items measure parent-child conflicts
Kessler Scale-6 | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  Screening for depression and anxiety the past 6 months
ISI-A | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  Form for assessing sleep disorders in children and adolescents
GTP-5 | Data will be collected at two time points; directly after the fourth and final treatment session and three months after completed treatment.
  Form for assessing gaming transfer phenomena

CONTACTS AND LOCATIONS:
Overall Officials: Emma Claesdotter-Knutsson, MD, PhD, Principal Investigator — Region Skane University Hospital, Lund University
Locations (1):
- BUP; Region Skane, Lund, Lund, Sweden

REFERENCES:
- [Derived] Werner M, Kapetanovic S, Claesdotter-Knutsson E. Family-Centered Treatment Program for Problematic Gaming and Excessive Screen Use in a Clinical Child and Youth Population (FAME): Protocol for a Feasibility Pilot Mixed Method Study. JMIR Res Protoc. 2024 Oct 8;13:e56387. doi: 10.2196/56387. PMID 39378066